CLINICAL TRIAL: NCT07169318
Title: A First-in-Human, 2-Part, Randomized, Double-Blind, Placebo-Controlled, Single Ascending Dose, Multiple Ascending Dose, and Food-Effect Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of VNT-101 Administered Orally to Healthy Adult Participants
Brief Title: First-in-Human Study of VNT-101: Safety, Tolerability, and Pharmacokinetics
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 23-0024; 75N93024F00001
Record Dates: First submitted 2025-07-03; First posted 2025-09-11 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2025-09-05

CONDITIONS: Influenza
Keywords: Double-Blind; First-in-Human; Food-Effect Study; Influenza; Multiple Ascending Dose; Nucleoprotein; Placebo-Controlled; Randomized; Safety; Single Ascending Dose; vnt-101
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: For both parts of the study, participants and the clinical personnel involved in the collection, monitoring, revision, or evaluation of AEs, or personnel who could have an impact on the outcome of the study will be blinded with respect to the participant's treatment assignment (VNT-101 or placebo)
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (18):
- Part 1 (SAD) Cohort S1 Arm 1 (Experimental): Healthy adult participants >/= 18 to 59 years will receive a Single Ascending Dose (SAD) of VNT-101 at 100 mg administered orally with approximately 240ml of water under fasting conditions. N=6
  Interventions: Drug: VNT-101
- Part 1 (SAD) Cohort S1 Arm 2 (Placebo Comparator): Healthy adult participants >/= 18 to 59 years will receive a Single Ascending Dose (SAD) of Placebo for VNT-101 at 100mg administered orally with approximately 240ml of water under fasting conditions. N=2
  Interventions: Other: Placebo for VNT-101
- Part 1 (SAD) Cohort S2 Arm 1 (Experimental): Healthy adult participants >/= 18 to 59 years will receive Single Ascending Dose (SAD) of VNT-101 at 250 mg administered orally with approximately 240ml of water under fasting conditions. N=6
  Interventions: Drug: VNT-101
- Part 1 (SAD) Cohort S2 Arm 2 (Placebo Comparator): Healthy adult participants >/= 18 to 59 years will receive a Single Ascending Dose (SAD) of Placebo for VNT-101 at 250mg administered orally with approximately 240ml of water under fasting conditions. N=2
  Interventions: Other: Placebo for VNT-101
- Part 1 (SAD) Cohort S3 Arm 1 (Experimental): Healthy adult participants >/= 18 to 59 years will receive a Single Ascending Dose (SAD) of VNT-101 at 500 mg administered orally with approximately 240ml of water under fasting conditions. N=6
  Interventions: Drug: VNT-101
- Part 1 (SAD) Cohort S3 Arm 2 (Placebo Comparator): Healthy adult participants >/= 18 to 59 years will receive a Single Ascending Dose (SAD) of Placebo for VNT-101 at 500mg administered orally with approximately 240ml of water under fasting conditions. N=2
  Interventions: Other: Placebo for VNT-101
- Part 1 (SAD) Cohort S4 Arm 1 (Experimental): Healthy adult participants >/= 18 to 59 years will receive a Single Ascending Dose (SAD) of VNT-101 at 1000 mg administered orally with approximately 240ml of water under fasting conditions. N=6
  Interventions: Drug: VNT-101
- Part 1 (SAD) Cohort S4 Arm 2 (Placebo Comparator): Healthy adult participants >/= 18 to 59 years will receive Single Ascending Dose (SAD) of Placebo for VNT-101 at 1000mg administered orally with approximately 240ml of water under fasting conditions. N=2
  Interventions: Other: Placebo for VNT-101
- Part 1 (SAD) Cohort S5 Arm 1 (Experimental): Healthy adult participants >/= 18 to 59 years from Cohort S3 will receive a Single Ascending Dose (SAD) of VNT-101 at 500 mg administered orally with approximately 240ml of water under fed (high-fat meal) conditions. N=6
  Interventions: Drug: VNT-101
- Part 1 (SAD) Cohort S5 Arm 2 (Placebo Comparator): Healthy adult participants >/= 18 to 59 years from Cohort 3 will receive a Single Ascending Dose (SAD) of Placebo for VNT-101 at 500mg administered orally with approximately 240ml of water under fed (high-fat meal) conditions. N=2
  Interventions: Other: Placebo for VNT-101
- Part 1 (SAD) Cohort S6 Arm 1 (Experimental): Healthy adult participants >/= 18 to 59 years will receive a Single Ascending Dose (SAD) of VNT-101 at 1500 mg administered orally with approximately 240ml of water under fasting conditions. N=6
  Interventions: Drug: VNT-101
- Part 1 (SAD) Cohort S6 Arm 2 (Placebo Comparator): Healthy adult participants >/= 18 to 59 years will receive a Single Ascending Dose (SAD) of Placebo for VNT-101 at 1500mg administered orally with approximately 240ml of water under fasting conditions. N=2
  Interventions: Other: Placebo for VNT-101
- Part 2 (MAD) Cohort M1 Arm 1 (Experimental): Following Single Ascending Dose (SAD) safety and Pharmacokinetics (PK) data review by the Safety Monitoring Committee (SMC), healthy adult participants >/= 18 to 59 years will receive Multiple Ascending Dose (MAD) of 250 mg of VNT-101 twice daily (BID) on Days 1 through 5 and 500mg of VNT-101 once daily (QD) on Day 6 administered orally with approximately 240ml of water under fasting conditions. N=8
  Interventions: Drug: VNT-101
- Part 2 (MAD) Cohort M1 Arm 2 (Placebo Comparator): Following Single Ascending Dose (SAD) safety and Pharmacokinetics (PK) data review by the Safety Monitoring Committee (SMC), healthy adult participants >/= 18 to 59 years will receive Multiple Ascending Dose (MAD) of 250 mg of Placebo for VNT-101 twice daily (BID) on Days 1 through 5 and 500mg of Placebo for VNT-101 once daily (QD) on Day 6 administered orally with approximately 240ml of water under fasting conditions. N=2
  Interventions: Other: Placebo for VNT-101
- Part 2 (MAD) Cohort M2 Arm 1 (Experimental): Following Single Ascending Dose (SAD) safety and PK data review by the Safety Monitoring Committee (SMC), healthy adult participants >/= 18 to 59 years will receive Multiple Ascending Dose (MAD) of 500 mg of VNT-101 twice daily (BID) on Days 1 through 5 and 1000mg of VNT-101 once daily (QD) on Day 6 administered orally with approximately 240ml of water under fasting conditions. N=8
  Interventions: Drug: VNT-101
- Part 2 (MAD) Cohort M2 Arm 2 (Placebo Comparator): Following Single Ascending Dose (SAD) safety and Pharmacokinetics (PK) data review by the Safety Monitoring Committee (SMC), healthy adult participants >/= 18 to 59 years will receive Multiple Ascending Dose (MAD) of 500 mg of Placebo for VNT-101 twice daily (BID) on Days 1 through 5 and 1000mg of Placebo for VNT-101 once daily (QD) on Day 6 administered orally with approximately 240ml of water under fasting conditions. N=2
  Interventions: Other: Placebo for VNT-101
- Part 2 (MAD) Cohort M3 Arm 1 (Experimental): Following Single Ascending Dose (SAD) safety and PK data review by the Safety Monitoring Committee (SMC), healthy adult participants >/= 18 to 59 years will receive Multiple Ascending Dose (MAD) of 750 mg of VNT-101 twice daily (BID) on Days 1 through 5 and 1500mg of VNT-101 once daily (QD) on Day 6 administered orally with approximately 240ml of water under fasting conditions. N=8
  Interventions: Drug: VNT-101
- Part 2 (MAD) Cohort M3 Arm 2 (Placebo Comparator): Following Single Ascending Dose (SAD) safety and Pharmacokinetics (PK) data review by the Safety Monitoring Committee (SMC), healthy adult participants >/= 18 to 59 years will receive Multiple Ascending Dose (MAD) of 750 mg of Placebo for VNT-101 twice daily (BID) on Days 1 through 5 and 1500mg of Placebo for VNT-101 once daily (QD) on Day 6 administered orally with approximately 240ml of water under fasting conditions. N=2
  Interventions: Other: Placebo for VNT-101

INTERVENTIONS:
Other: Placebo for VNT-101 — Capsules will be size 00 and filled with microcrystalline cellulose
  Arms: Part 1 (SAD) Cohort S1 Arm 2; Part 1 (SAD) Cohort S2 Arm 2; Part 1 (SAD) Cohort S3 Arm 2; Part 1 (SAD) Cohort S4 Arm 2; Part 1 (SAD) Cohort S5 Arm 2; Part 1 (SAD) Cohort S6 Arm 2; Part 2 (MAD) Cohort M1 Arm 2; Part 2 (MAD) Cohort M2 Arm 2; Part 2 (MAD) Cohort M3 Arm 2
Drug: VNT-101 — VNT-101 is an orally bioavailable, direct-acting antiviral with a novel mechanism of action - inhibiting oligomerization of the influenza nucleoprotein (NP) and thereby inhibiting viral ribonucleic acid (RNA) synthesis.
  Arms: Part 1 (SAD) Cohort S1 Arm 1; Part 1 (SAD) Cohort S2 Arm 1; Part 1 (SAD) Cohort S3 Arm 1; Part 1 (SAD) Cohort S4 Arm 1; Part 1 (SAD) Cohort S5 Arm 1; Part 1 (SAD) Cohort S6 Arm 1; Part 2 (MAD) Cohort M1 Arm 1; Part 2 (MAD) Cohort M2 Arm 1; Part 2 (MAD) Cohort M3 Arm 1

SUMMARY:
A randomized, double-blind, placebo-controlled Phase 1 study conducted at a single center with approximately 78 healthy adults aged 18-59 years. Part 1 Single Ascending Dose (SAD) will enroll 48 participants into six cohorts (S1-S6) to receive single oral doses of VNT-101 (100-1500 mg) or placebo under fasting or fed (S5 only) conditions. Part 2 Multiple Ascending Dose (MAD) will enroll 30 participants into three cohorts (M1-M3) to receive multiple oral doses of VNT-101 (250-750 mg BID Days 1-5, QD Day 6) or placebo under fasting conditions. Dose escalation in both parts will proceed after Protocol Safety Review Team (PSRT) review. The primary objective for Part 1 is to evaluate the safety and tolerability of single ascending oral (SAD) doses of VNT-101 in healthy adult participants under either fasting or fed conditions. The primary objective for part 2 is to evaluate the safety and tolerability of multiple ascending oral (MAD) doses of VNT-101 in healthy adult participants.

DETAILED DESCRIPTION:
This will be a single center, Phase 1, placebo-controlled, randomized, double-blind, integrated sequential Single Ascending Dose (SAD) (with a food-effect cohort) and Multiple Ascending Dose (MAD) study. The study will be divided into two parts, Part 1: SAD cohorts, with a cohort for food effect evaluation and Part 2: MAD cohorts. Part 1 will be completed sequentially with Protocol Safety Review Team (PSRT) reviews before advancing to the next higher dose. An interim analysis will be performed and reviewed by the SMC before the start of Part 2 and complete ascending dose levels sequentially.

Part 1 will consist of 6 cohorts (1 cohort per dose level). Approximately 48 healthy adult participants in 6 cohorts (S1 to S6) are planned for sequential randomization and evaluation. Each cohort will include 8 participants (6 participants will be administered the study product VNT-101 and 2 matching placebo). SAD doses planned of VNT-101 range from a starting dose of 100 mg up to a highest dose of 1500 mg. Cohorts S1, S2, S3, S4, and S6 will be dosed in a double-blinded manner in a fasting state, whereas Cohort S5 will be dosed in a blinded manner in the fed state (high-fat meal) and will consist of the 8 participants who participated in Cohort S3, showing AUC and Cmax exposures at least 3-fold less than the cohort dose escalation criteria for exposure limit for AUD and Cmax. If AUC or Cmax are within 3-fold of the halting limit, then Cohort S5 may utilize the lower dose of 250mg evaluated in participants from Cohort S2, who were given a lower dose of 250mg in the fasted state, unless the PSRT decides a different cohort (Cohort S2) should return based on blinded Pharmacokinetics (PK) results. The primary objective for Part 1 is to evaluate the safety and tolerability of single ascending oral (SAD) doses of VNT-101 in healthy adult participants under either fasting or fed conditions. The secondary objective of part 1 is to characterize the PK profile of VNT-101 in plasma after single oral dose of VNT-101 in fasted healthy adult participants and one dose in fed healthy adult participants.

In Part 2, approximately 30 healthy adult participants in 3 cohorts (Cohorts M1 to M3) of 10 participants each (8 active and 2 placebo) are planned for sequential randomization and evaluation. Cohorts will be dosed sequentially in an ascending fashion. In each cohort, participants will receive under fasting conditions 11 oral doses of VNT-101 or placebo twice daily (BID) for 5 days with an additional dose being administered on the morning of Day 6. The primary objective for part 2 is to evaluate the safety and tolerability of multiple ascending oral (MAD) doses of VNT-101 in healthy adult participants. The Secondary objectives are 1) To characterize the PK profile of VNT-101 in plasma after multiple oral doses of VNT-101 in healthy adult participants and 2) To characterize the PK profile of VNT-101 in urine after multiple oral doses of VNT-101 in healthy adult participants.

ELIGIBILITY:
Inclusion Criteria:

1. Provides written informed consent prior to the initiation of any trial procedures.
2. Able to understand and agrees to comply with all planned trial procedures and be available for all study visits.
3. Healthy, adult, male or female (of non-childbearing potential only*), 18-59 years of age, inclusive, at the screening visit.

   * Female participants of non-childbearing potential must be either surgically sterile (i.e., hysterectomy, bilateral tubal ligation, bilateral tubal occlusion [hysteroscopic sterilization], salpingectomy, and/or bilateral oophorectomy at least 26 weeks before Screening) or post-menopausal, defined as spontaneous amenorrhea for at least a year, with follicle-stimulating hormone (FSH) in the post-menopausal range at Screening, based on the central laboratory ranges.
4. Continuous non-smoker who has not used nicotine-, tobacco-, cannabis-, or cannabidiol-containing products** prior to the first dosing based on participant self-reporting.

   **The period before first dose is at least 3 months for tobacco and associated products and at least 60 days for cannabis and associated products.
5. Body mass index (BMI)>/=18.0 and </= 30.0 kg/m^2 at the screening visit.
6. Medically healthy*** with no clinically significant medical history, physical examination, laboratory profiles, vital signs, and ECGs, as deemed by the Principal Investigator (PI) or designee,

   ***Including the following:
   1. Supine diastolic blood pressure is >/= 40 mmHg and </= 90 mmHg at the screening visit.
   2. Supine systolic blood pressure is >/= 90 mmHg and </= 140 mmHg at the screening visit.
   3. Supine heart rate is >/= 60 bpm and</= 100 bpm at the screening visit.
   4. QTcF interval is </= 460 msec (males) and </=470 msec (females) and has ECG findings considered normal or not clinically significant by the PI or designee at the screening visit.
   5. Estimated creatinine clearance >/= 80 mL/min based on the Cockroft-Gault equation and creatinine <1.50 mg/dL at the screening visit.
   6. Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) is not greater than 1.1 times the upper limit of normal (ULN), as specified by the testing laboratory.
   7. Other clinical laboratory values within normal range as specified by the testing laboratory, unless deemed not clinically significant by the PI or designee.
7. Must agree to refrain from using tanning salons, saunas, sunbathing, or prolonged sun exposure during participation in the study through the follow-up visit.
8. Male participants must agree not to donate sperm during the study and for 90 days following the last administration of Study Product.
9. Male participants must agree to use a medically accepted contraceptive regimen**** during participation and for 30 days after last administration of the study product or be vasectomized.

   * Acceptable methods of contraception include abstinence from intercourse with a female of childbearing potential or use of male condoms with spermicide or surgical sterilization (vasectomy) of participant at least 26 weeks before the Screening.

Exclusion Criteria:

1. History or presence of clinically significant medical or psychiatric condition or disease, making the participant unsuitable for enrollment in the opinion of the PI or designee.
2. History of severe allergic or anaphylactic reactions to any prescription or non-prescription drug or vaccine.
3. Participants who took any prescription medications within 14 days of first dosing or within 5 half-lives of the drug, whichever is longer.
4. Participants who took any over the counter (OTC) medication/vitamins/herbal supplements* in the last 7 days prior to first dosing.

   *Exception for occasional use of OTC acetaminophen (paracetamol) 325 to 500 mg every 4 hours not to exceed 3000 mg/day.
5. History or diagnosis of a cardiovascular disease condition, including myocardial infarction, angina, congenital heart disease, cardiomyopathy, hypertension, or hypercholesteremia**.

   **Defined as: clinically significant hypercholesteremia with high low-density lipoprotein (LDL) cholesterol (>/= 160 mg/dL)
6. Increased risk for peptic ulcer***

   ***Defined as: participants with a history of gastric or duodenal ulcer, chronic non-steroidal anti-inflammatory drug use in the past 3 months, current smokers, alcohol consumption of > 21 alcoholic units per week (where 1 unit = 284 mL of beer, 25 mL of 40% spirit or a 125 mL of wine) or chronic atrophic gastritis,
7. Female participant with a positive pregnancy test at the screening visit or at baseline or who is lactating.
8. Positive urine drug toxicology test (or cotinine or alcohol results) at the screening visit or check-in.
9. Has been on a diet incompatible with the on-study diet****, in the opinion of the PI or designee, within the 30 days prior to the first dosing,

   ****including consumption of grapefruit/Seville orange within 14 days prior to first dosing,
10. For Cohorts S2, S3, and S5 only, is known to be intolerant of a high fat/high calorie diet.
11. Participants who are unlikely to comply with the study protocol OR those who would not be suitable candidates for participation in the opinion of the investigator.
12. Participants who donated blood or plasma recently*****

    *****Recently defined as within 30 days prior to Day -1, or loss of whole blood of more than 500 mL within 30 days prior to Day-1, or receipt of a blood transfusion within 1 year of study enrollment.
13. Participated in a clinical study involving administration of an investigational drug in the past 30 days (90 days for injectable biological agent) before screening.

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 78 (Estimated)
Dates: Start 2025-09-16 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Change from baseline blood pressure (BP) | Day 1 through Day 13
Change from baseline heart rate (HR) | Day 1 through Day 13
Change from baseline heart rhythm, measured by a 12-lead safety Electrocardiogram (ECG) | Day 1 through Day 13
  12-lead ECG will be measured in triplicate
Change from baseline Hemoglobin | Day 1 through Day 8
Change from baseline in Absolute neutrophil count | Day 1 through Day 13
Change from baseline in active partial thromboplastin time | Day 1 through Day 13
Change from baseline in blood in urine | Day 1 through Day 13
Change from baseline in direct serum Bilirubin | Day 1 through Day 13
Change from baseline in Hematocrit | Day 1 through Day 13
Change from baseline in international normalized ratio | Day 1 through Day 13
Change from baseline in lipase in Single Ascending Dose (SAD) | Day 1 through Day 13
Change from baseline in prothrombin time | Day 1 through Day 13
Change from baseline in red blood cell count | Day 1 through Day 13
Change from baseline in serum Alanine aminotransferase | Day 1 through Day 13
Change from baseline in serum Albumin | Day 1 through Day 13
Change from baseline in serum Alkaline phosphatase | Day 1 through Day 13
Change from baseline in serum Aspartate Aminotransferase | Day 1 through Day 13
Change from baseline in serum Bicarbonate | Day 1 through Day 13
Change from baseline in serum Blood Urea Nitrogen | Day 1 through Day 13
Change from baseline in serum Chloride | Day 1 through Day 13
Change from baseline in serum Creatinine | Day 1 through Day 13
Change from baseline in serum Glucose | Day 1 through Day 13
Change from baseline in serum Potassium | Day 1 through Day 13
Change from baseline in serum Sodium | Day 1 through Day 13
Change from baseline in total serum Bilirubin | Day 1 through Day 13
Change from baseline in urine leukocyte esterase | Day 1 through Day 13
Change from baseline in urine nitrate level | Day 1 through Day 13
Change from baseline in urine protein | Day 1 through Day 13
Change from baseline in White blood cell count with differential | Day 1 through Day 13
Change from baseline oral temperature | Day 1 through Day 13
Change from baseline Platelet count | Day 1 through Day 13
Change from baseline PR interval, measured by a 12-lead safety Electrocardiogram (ECG) | Day 1 through Day 13
  12-lead ECG will be measured in triplicate
Change from baseline QRS duration, measured by a 12-lead safety Electrocardiogram (ECG) | Day 1 through Day 13
  12-lead ECG will be measured in triplicate
Change from baseline QT interval, measured by a 12-lead safety Electrocardiogram (ECG) | Day 1 through Day 13
  12-lead ECG will be measured in triplicate
Change from baseline QTcF interval, measured by a 12-lead safety Electrocardiogram (ECG) | Day 1 through Day 13
  12-lead ECG will be measured in triplicate
Change from baseline respiratory rate (RR) | Day 1 through Day 13
Change from baseline RR interval, measured by a 12-lead safety Electrocardiogram (ECG) | Day 1 through Day 13
  12-lead ECG will be measured in triplicate
Incidence of Treatment Emergent Adverse Events (TEAEs) | Day 1 through Day 13
Proportion of participants with findings from cardiac telemetry | Day 1 through Day 13
  Cardiac telemetry will monitor heart rate and rhythm
Proportion of participants with findings from physical examination. | Day 1 through Day 8
Proportion of participants with findings from visual exam of clean-catch urine sample | Day 1 through Day 13

SECONDARY OUTCOMES:
Accumulation ratio based on area under the concentration curve (RA_AUC) in plasma | Through Day 9
  Multiple Ascending Dose (MAD) cohorts only.
Accumulation ratio based on Cmax (RA_Cmax) in plasma | Through Day 9
  Multiple Ascending Dose (MAD) cohorts only.
Amount of drug excreted unchanged between t1 and t2 (Aet1-t2,ss) in urine | Through Day 9
  Multiple Ascending Dose (MAD) cohorts only.
Apparent volume of distribution at terminal phase (VZ/F) in plasma | Day 1 through Day 4
  Single Ascending Dose (SAD) cohorts only.
Apparent volume of distribution at terminal phase at a steady state (Vz,ss/F) in plasma | Through Day 9
  Multiple Ascending Dose (MAD) cohorts only.
Area under the concentration curve from time 0 to 12 hours (AUC0-12) in plasma | Day 1 through Day 9
Area under the concentration curve from time 0 to infinity (AUC0-infinity) in plasma | Day 1 through Day 4
  Single Ascending Dose (SAD) cohorts only.
Area under the concentration curve from time 0 to time t (AUC0-t) in plasma | Day 1 through Day 9
Area under the concentration versus time curve over the dosing interval, tau (AUCtau) in plasma | Through Day 9
  Multiple Ascending Dose (MAD) cohorts only.
Calculated average concentration (Cavg) in plasma | Through Day 9
  Multiple Ascending Dose (MAD) cohorts only.
Change from baseline in clearance at a steady state (CLss/F) in plasma | Through Day 9
  Multiple Ascending Dose (MAD) cohorts only.
Clearance (CL/F) in plasma | Day 1 through Day 4
  Single Ascending Dose (SAD) cohorts only.
Cumulative amount of drug excreted unchanged (CumAess) in urine | Through Day 9
  Multiple Ascending Dose (MAD) cohorts only.
Cumulative fraction of drug excreted unchanged (CumFess) in urine | Through Day 9
  Multiple Ascending Dose (MAD) cohorts only.
Elimination half-life (t1/2) in plasma | Day 1 through Day 9
Fraction of drug excreted unchanged between t1 and t2 (Fet1-t2,ss) in urine | Through Day 9
  Multiple Ascending Dose (MAD) cohorts only.
Maximum observed concentration (Cmax) in plasma | Day 1 through Day 9
Maximum observed concentration (Ctrough) in plasma | Through Day 9
  Multiple Ascending Dose (MAD) cohorts only.
Maximum observed plasma concentration at a steady state (Cmax,ss) in plasma | Through Day 9
  Multiple Ascending Dose (MAD) cohorts only.
Minimum observed plasma concentration at a steady state (Cmin,ss) in plasma | Through Day 9
  Multiple Ascending Dose (MAD) cohorts only.
Renal clearance at steady state (CLrss) | Through Day 9
  Multiple Ascending Dose (MAD) cohorts only.
Terminal elimination rate constant (Kel) in plasma | Day 1 through Day 9
Time of observed maximum concentration (Tmax) at a steady state (Tmax,ss) in plasma | Through Day 9
  Multiple Ascending Dose (MAD) cohorts only.

CONTACTS AND LOCATIONS:
Locations (1):
- Altasciences Inc - Kansas City, Overland Park, Kansas, United States